CLINICAL TRIAL: NCT07225140
Title: A Multicenter, Double-blind, Randomized, Parallel Group, Active-controlled, Dose-ranging Study to Assess Efficacy, Safety, and Pharmacokinetics of Combogesic® 325 in Adolescent Patients (Aged 12 to Less Than 18 Years) With Moderate to Severe Postoperative Pain Associated With Orthopedic Surgery
Brief Title: A Study of Combogesic® 325 in Adolescent Patients With Moderate to Severe Postoperative Pain Associated With Orthopedic Surgery
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AFT Pharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFT-MX-16p
Record Dates: First submitted 2025-10-30; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A- 3 tablets of Combogesic® tablets (Experimental): 3 tablets of Combogesic® (acetaminophen 975mg + ibuprofen 292.5 mg, total per dose) will be administered every 6 hours up to a maximum of 4 doses in 24 hours.
  Interventions: Drug: Combogesic® tablets
- Treatment B- 2 tablets of Combogesic® + 1 tablets of placebo (Experimental): 2 tablets of Combogesic® (acetaminophen 650 mg + ibuprofen 195 mg, total per dose) and 1 tablet of placebo will be administered every 6 hours up to a maximum of 4 doses in 24 hours.
  Interventions: Drug: Combogesic® tablets; Drug: Placebo
- Treatment C - 2 tablets of acetaminophen and 1 tablet of placebo (Active Comparator): 2 tablets of acetaminophen (1000 mg total per dose) + 1 tablet of placebo will be administered every 6 hours up to a maximum of 4 doses in 24 hours.
  Interventions: Drug: Acetaminophen 500mg; Drug: Placebo

INTERVENTIONS:
Drug: Combogesic® tablets — The active ingredients of Combogesic® tablets are acetaminophen 325 mg and ibuprofen 97.5 mg.
  Other Names: Acetaminophen 325 mg and ibuprofen 97.5 mg
  Arms: Treatment A- 3 tablets of Combogesic® tablets; Treatment B- 2 tablets of Combogesic® + 1 tablets of placebo
Drug: Acetaminophen 500mg — Each tablet contains acetaminophen 500mg.
  Arms: Treatment C - 2 tablets of acetaminophen and 1 tablet of placebo
Drug: Placebo — Placebo tablets do not contain any active ingredients
  Arms: Treatment B- 2 tablets of Combogesic® + 1 tablets of placebo; Treatment C - 2 tablets of acetaminophen and 1 tablet of placebo

SUMMARY:
Combogesic® 325 contains a combination of ibuprofen and acetaminophen. The purpose of this study is to compare the pain relief effects of Combogesic® 325mg and acetaminophen and to evaluate the safety of Combogesic® 325mg in adolescents between the ages of 12 and <18 years.

What will the study involve for participants?

* Participants will be randomly allocated to one of 3 treatment groups:

  * 3 tablets of Combogesic® 325,
  * 2 tablets of Combogesic® 325 and 1 tablet of placebo or
  * 2 tablets of acetaminophen1000mg and 1 tablet of placebo
* Participants will take 3 tablets every 6 hours with a maximum of 4 doses in 24 hours
* Participants and study doctor will be blinded to the treatment group
* If pain is not sufficiently controlled, opioids may be used as supplementary pain relief at the discretion of the study doctor.
* Participants will complete a patient diary to assess their pain
* Participants will rate the study drug at the end of the treatment.

It is expected that Combogesic® tablets (either 2 or 3 tablets per dose) will provide a greater reduction in pain compared to acetaminophen (1000 mg) treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent or consent be provided from parents/legal guardians and assent from participants (where appropriate).
* Be males and females aged at least 12 years and less than 18 years old on both the day of consent and throughout the 24 hour study period.
* Be undergoing planned orthopedic surgery which requires at least 24 hours of hospital inpatient stay.
* Have a clinical indication of acute moderate or severe pain (at least ≥ 50 mm on the VAS scale*) within 6 hours after the completion of surgery associated with orthopedic surgery.
* using a 100mm VAS scale with 0 = no pain and 100 = worst pain imaginable, patients should have a resting VAS pain intensity score of ≥ 50 mm for inclusion. For this study, moderate pain is defined as ≥ 40 mm to ≤ 69 mm and severe pain is defined as a resting VAS of ≥ 70 mm to ≤ 100 mm.
* Have negative HIV and hepatitis B & C test results.

Exclusion Criteria:

* Has taken any NSAID or acetaminophen containing drug products within 5 half-lives prior to the initial dose of study drug.
* Hypersensitivity to opioids, NSAIDs or acetaminophen or a history of severe/serious drug reaction to NSAIDs or acetaminophen.
* Pregnant or lactating females Known to be pregnant or possibly pregnant.
* Sexually active females of childbearing potential not using adequate contraception* and sexually active males not using adequate contraception**
* Women of childbearing potential who are unwilling to take adequate contraceptive precautions, i.e., a hormonal contraceptive, an intrauterine device, double-barrier method, or abstinence (should the participant become sexually active, she must agree to use a double-barrier method of contraception). A woman of childbearing potential is defined as any female who is less than 2 years post-menopausal or has not undergone a partial or total hysterectomy or surgical sterilization, e.g. bilateral tubal ligation, bilateral oophorectomy.
* Women of childbearing potential who are unwilling to undergo a urine pregnancy test.
* Suffering from a neurological disorder relating to pain perception or any acute or chronic condition that, in the opinion of the Investigator, makes the participant unsuitable from an efficacy or safety perspective.
* In the opinion of the Investigator, unable to understand the visual analogue pain score or comply with the protocol requirements.
* Currently or in last 30 days, has been in a clinical trial involving another study drug.
* Have donated blood or blood products within 30 days prior to study drug administration
* Advanced renal impairment (serum creatinine >132 µmol/L) or a risk for renal failure due to volume depletion.
* Severe known haemopoietic, renal or hepatic disease, or immunosuppressed, including any clinically significant finding from the laboratory tests results (biochemistry and hematology at screening), which, in the opinion of the Investigator, means that it would not be in the participants' best interests to participate in this study.
* History of gastric ulceration or other GI disorders that, in the opinion of the Investigator make the participant unsuitable (e.g. frequent treatment of gastroesophageal reflux disease, inflammatory bowel disease, etc).
* History of severe asthma in the opinion of the investigator.
* Has a history of drug or alcohol abuse
* Suffering from any other disease or condition which, in the opinion of the Investigator, means that it would not be in the participant's best interests to participate in this study.

  * Methods of contraception that are deemed adequate have failure rates of < 1%, including: established use of oral contraceptives in conjunction with a barrier method of contraception; injected or implanted hormonal methods of contraception; placement of intrauterine device (IUD) or intrauterine system (IUS); sexual abstinence; hysterectomy; post-menopausal; sterilized; vasectomy. Suitable contraception should be used for the entire study period, from screening to follow-up. Women of childbearing age include all women that have begun puberty and had their first menstrual period until they reach menopause.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time-adjusted summed pain intensity difference (SPID) calculated from the visual analogue scale (VAS) pain intensity scores 6 hours after first dose of study medication | From start of exposure to study drug until 6 hours after first dose
  SPID will be derived from the 100 mm Visual Analogue Scale which is the tool used for patients to rate the intensity of their pain on a horizontal 100mm line with 0 on one end and 100 on the other end (0 being no pain and 100 being the worst pain unimaginable). The primary analysis will compare three tablets of Combogesic® against acetaminophen

SECONDARY OUTCOMES:
Time-adjusted SPID0-6 (for 2 tablets of Combogesic vs. acetaminophen) and Time-adjusted SPID0-12, SPID0-18 and SPID0-24 for both doses. | From start of exposure to study medication up to 24 hours
The time to onset of pain relief after the first dose of study drug defined as (i) perceptible, (ii) meaningful and (iii) complete pain relief using the three stopwatch method. | From start of exposure to study medication up to 24 hours
The maximum VAS pain scores up to 24 hours after the first dose of study medication. | From start of exposure to study medication up to 24 hours
  100 mm Visual Analogue Scale is the tool used for patients to rate the intensity of their pain on a horizontal 100mm line with 0 on one end and 100 on the other end (0 being no pain and 100 being the worst pain unimaginable)
The pain intensity (PI) and pain intensity difference (PID) at 6, 12, 18, and 24 hours after first dose. | From start of exposure to study medication up to 24 hours
  100 mm Visual Analogue Scale which is the tool used for patients to rate the intensity of their pain on a horizontal 100mm line with 0 on one end and 100 on the other end (0 being no pain and 100 being the worst pain unimaginable). The PID will be measured by the difference between the baseline score and the score at 6, 12, 18, and 24 hours after first dose.
Pain relief as measured on a 5-point categorical scale at 6, 12, 18, and 24 hours after first dose. | From start of exposure to study medication up to 24 hours
  Patients will be asked to rate their pain in their patient diary with the following questionnaire.
  Please rate your pain relief:
  0= no pain relief; (the pain is the same, or worse, than the starting pain)
  1. a little pain relief; (the pain is less than half gone)
  2. some pain relief; (the pain is about half gone)
  3. a lot of pain relief; (the pain is more than half gone)
  4. complete pain relief; (the pain is completely gone)
Peak pain relief | From start of exposure to study medication up to 24 hours
Time to peak pain relief | From start of exposure to study medication up to 24 hours
Total pain relief (TOTPAR) (calculated as a time-weighted average) over 0-6 hours (TOTPAR-6), over 0-12 hours (TOTPAR-12), over 0-18 hours (TOTPAR-18), and over 0-24 hours (TOTPAR-24). | From start of exposure to study medication up to 24 hours
The response rates (response rate to be defined as the percentage of participants who reduce their pain intensity scores by at least 50% compared with the baseline VAS measure). | From start of exposure to study medication up to 24 hours
Time to response | From start of exposure to study medication up to 24 hours
The time to requirement for rescue medication. | From start of exposure to study medication up to 24 hours
The percentage of participants using rescue medication at 6, 12, 18, and 24 hours after first dose. | From start of exposure to study medication up to 24 hours
Total Dose (mg) of primary (oxycodone) and secondary (morphine) rescue medication over 24 hours | From start of exposure to study medication up to 24 hours
Total oral Morphine Milligram Equivalent (MME) dose of all rescue medication over the 24 hour study period | From start of exposure to study medication up to 24 hours
The categorical global evaluation of study drug. | From start of exposure to study medication up to 24 hours
  Each patient will rate the study medication using a questionnaire of: How do you rate the study medication? 1 = Poor; 2 = Fair; 3 = Good; 4 = Very Good; 5 = Excellent The patient's global evaluation of the study drug will be summarized by the number and percentage of subjects within each category.
To compare treatment-emergent adverse event (TEAE) rates over the course of treatment and at a follow up call 7 days after last dose. | From start of exposure to study medication until 7 days after last dose
The incidence of specific NSAID and acetaminophen adverse effects from the first dose of study drug until Day 7. | From start of exposure to study medication until 7 days after final dose
  Adverse effects include GI ulceration or bleeding, indigestion/stomach pain, post-operative bleeding, bronchospasm, skin reactions, water retention, renal failure, thromboembolic events, and evidence of clinical hepatitis
To characterize the pharmacokinetic profile of two different doses of Combogesic® 325 (T1/2- Time required for the plasma drug concentration to decrease by one half) | Approximately 15 minutes before first dose of study medication until 6 hours after first study medication administration and before second dose
  This will be defined from the plasma concentration versus time data using non-compartmental methods
To characterize the pharmacokinetic profile of two different doses of Combogesic® 325 (Extrapolated AUC(0-∞)- The area under the plasma concentration versus time curve, from zero to infinity) | Approximately 15 minutes before first dose of study medication until 6 hours after first study medication administration and before second dose
  This will be defined from the plasma concentration versus time data using non-compartmental methods
To characterize the pharmacokinetic profile of two different doses of Combogesic® 325 (Cmax- Maximum measured plasma concentration) | Approximately 15 minutes before first dose of study medication until 6 hours after first study medication administration and before second dose
  This will be defined from the plasma concentration versus time data using non-compartmental methods
To characterize the pharmacokinetic profile of two different doses of Combogesic® 325 (Tmax- Time to maximum measured plasma concentration) | Approximately 15 minutes before first dose of study medication until 6 hours after first study medication administration and before second dose
  This will be defined from the plasma concentration versus time data using non-compartmental methods
To characterize the pharmacokinetic profile of two different doses of Combogesic® 325 (AUC(0-t) - The area under the plasma concentration versus time curve from time zero to the last measurable concentration) | Approximately 15 minutes before first dose of study medication until 6 hours after first study medication administration and before second dose
  This will be defined from the plasma concentration versus time data using non-compartmental methods

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Health, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No